CLINICAL TRIAL: NCT00305058
Title: A Randomized Clinical Trial Comparing Intravenous Morphine and Intravenous Hydromorphone in the Treatment of Adult ED Patients With Moderate to Severe Pain
Brief Title: Trial Comparing Morphine to Hydromorphone in Elderly Patients With Severe Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, Assistant Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMC 04-08-225E
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Acute Pain
Keywords: Elderly; Hydromorphone; Morphine; Pain; Acute; Emergency Department
MeSH Terms: conditions — Acute Pain; Pain; Emergencies | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Hydromorphone (Experimental): 0.0075 mg/kg IV hydromorphone
  Interventions: Drug: Hydromorphone
- Morphine (Active Comparator): 0.05 mg/kg IV morphine
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — 0.05 mg/kg Intravenous
  Arms: Morphine
Drug: Hydromorphone — 0.0075 mg/kg intravenous
  Other Names: Dilaudid
  Arms: Hydromorphone

SUMMARY:
The purpose of this research study is to determine which opiate pain medication (morphine or hydromorphone (Dilaudid)) is more effective in the treatment of acute pain in patients presenting to the emergency department.

DETAILED DESCRIPTION:
Pain is cited as the most frequent reason for visit to emergency departments (EDs) . It can be estimated from the National Hospital Ambulatory Medical Care Survey, an annual survey of a representative sample of visits to US EDs, that there are 17 million visits per year to US EDs for specific complaints of pain, 29 million visits including "back symptoms" and "injuries not otherwise specified" as well as specific mentions of pain. However it is widely acknowledged that pain is seriously under-treated in the ED as well as in other health care settings. The concern regarding under-treatment is reflected in new standards for pain management developed by the Joint Commission on Accreditation of Healthcare Organizations (JCAHO) requiring assessment of pain at triage in the ED and referring to pain measurement as the "fifth vital sign".

Proper pain management is a tremendous challenge to ED physicians as pain is not only a noxious experience but also a symptom of injury and disease that needs to be understood and appropriately treated. Further complicating pain management is the large interpersonal variability in pain perception and expression reflecting cultural, contextual, and individual differences between people. Reasons for under-treating pain include concern over side effects of opioids, perception of pain complaints as possible drug-seeking behavior, under-staffing, concern that analgesics will mask symptoms, delay early diagnosis, treatment, and contribute to risks of tolerance and dependence in vulnerable patients.

The elderly represent a group of patients who may experience pain differently from the non-elderly patient. This growing population has been significantly underrepresented in pain-related studies. Some studies have shown that the elderly are at risk for "oligoanalgesia" and receive inadequate doses of pain medication.

Morphine has long been considered the gold standard in pain control. Hydromorphone is another powerful opiate that has been used extensively for the management of post-operative pain and morphine-resistant cancer-related pain. A recent Cochrane review on the use of hydromorphone found 32 studies that focused on acute pain. Of these 32 studies, only 9 involved intravenous forms of hydromorphone. Of these 8 studies, 5 involved patient controlled analgesia, and only 1 study compared intravenous (IV) hydromorphone to IV morphine. The Cochrane review concludes that there are gaps in the understanding of the efficacy and potency of hydromorphone. Only 1 study of hydromorphone in the ED could be located and this compared IV hydromorphone versus IV meperidine in patients with ureteral colic. Although this study showed hydromorphone was superior at all time periods and had fewer side effects, the study used fixed doses of hydromorphone (1mg) and meperidine (50mg).

It has been the clinical experience of some ED physicians that hydromorphone may be a better opiate in patients presenting to the ED with acute pain. Hydromorphone is also the opiate that is usually given if morphine does not adequately control a patient's pain in the ED.

Hydromorphone may also have other benefits, such as a faster onset since it is more lipophilic than morphine and crosses the blood-brain barrier faster.

If it is shown that hydromorphone gives better pain relief to patients with comparable or fewer side effects when compared with morphine, then we may be able to provide evidence to suggest that hydromorphone should be the parenteral opiate of choice for adult ED patients presenting with acute pain of moderate to severe intensity.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 65 years
2. Pain with onset within 7 days
3. ED attending physician's judgment that patient's pain warrants use of parenteral opioids
4. Normal mental status

Exclusion Criteria:

1. Prior use of methadone
2. Use of other opioids or tramadol within past seven days
3. Prior adverse reaction to morphine or hydromorphone
4. Chronic pain syndrome
5. Alcohol intoxication
6. Systolic Blood Pressure <90 mm Hg
7. Use of monoamine oxidase (MAO) inhibitors in past 30 days
8. Elderly patients with a capnometry reading of greater than 46

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 194 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew K Chang, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morphine | Hydromorphone
Started | 97 | 97
Inclusion/Exclusion Verification | 96 | 97
All Outcome Data Collected | 93 | 95
Data Collection Forms Filed for Analysis | 90 | 93
Completed | 90 | 93
Not Completed | 7 | 4
Not completed — Participant too young | 1 | 0
Not completed — Missing data collection instrument | 3 | 2
Not completed — Missing outcome data | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Hydromorphone | Total
Number analyzed (Participants) | 90 | 93 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (8) | 74 (8) | 75 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 65 | 128
  Male | 27 | 28 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 39 | 47 | 86
  Black | 21 | 28 | 49
  White | 27 | 18 | 45
  Other | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90 | 93 | 183
Weight [Mean (Standard Deviation); unit: lbs] | 148 (29) | 157 (29) | 153 (29)
Primary Language [Count of Participants; unit: Participants]
  English | 51 | 51 | 102
  Spanish | 33 | 40 | 73
  Other | 5 | 0 | 5
  Unknown | 1 | 2 | 3
Baseline Pain Score [Count of Participants; unit: Participants] — based on a numerical rating scale (NRS) of 0 ("no pain") to 10 ("worst possible pain")
  Participants
    6 | 9 | 10 | 19
    7 | 12 | 9 | 21
    8 | 20 | 18 | 38
    9 | 9 | 10 | 19
    10 | 40 | 46 | 86
Number of participants who took analgesics before coming to the ED [Count of Participants; unit: Participants]
  None | 66 | 75 | 141
  Some | 24 | 18 | 42
Number of participants who had pain in specific locations [Count of Participants; unit: Participants]
  Abdomen/pelvis | 45 | 56 | 101
  Extremities | 5 | 8 | 13
  Back | 18 | 7 | 25
  Chest | 2 | 4 | 6
  Head/neck | 2 | 2 | 4
  Other | 18 | 15 | 33
  Unknown/missing data | 0 | 1 | 1
Number of participants experiencing nausea since pain began [Count of Participants; unit: Participants]
  No | 48 | 48 | 96
  Yes | 41 | 38 | 79
Number of participants experiencing vomiting since pain began [Count of Participants; unit: Participants]
  No | 59 | 60 | 119
  Yes | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: Pain scores are a measure of pain intensity and are measured on the numerical rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable). Participants are asked to rate their pain using this scale at baseline before any medication is administered and again 30 minutes after medication is infused
Time Frame: Baseline to 30 minutes after medication infused
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 90 | 93
units on a scale | 3.3 (2.5) | 3.8 (2.6)

2. Secondary Outcome: Number of Participants With a Change in Pain Score
Description: Pain score is a measure of pain intensity using the numerical rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable). Data is separated into two groups: those with greater than or equal to 50% change in their pain score and those with less than 50% change in their pain score.
Time Frame: Baseline to 30 minutes after medication infused
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 90 | 93
Participants
  less than 50% decrease | 53 | 53
  greater than or equal to 50% decrease | 37 | 40

3. Secondary Outcome: Number of Participants With Pain Relief
Description: Pain relief here is a subjective measure indicated by the following categories: No, Slight, Moderate, and Complete. Participants were asked to pick the category that best fit their level of pain relief 30 minutes after medication was infused.
Time Frame: 30 minutes after medication infused
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 90 | 93
Participants
  none or slight | 37 | 32
  moderate to complete | 53 | 61

4. Secondary Outcome: Number of Participants Satisfied With Pain Medication
Description: Number of participants who were satisfied with pain medication received, based on their response of good to excellent or poor to fair. Participants were asked to pick which response best fit their satisfaction with the pain medication they received 30 minutes after that medication was infused "Good to Excellent" or "Poor to fair".
Time Frame: 30 minutes after medication infused
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 90 | 93
Participants
  Good to excellent | 56 | 59
  Poor to fair | 34 | 34

ADVERSE EVENTS:
Time Frame: 120 minutes
Arm/Group | Morphine | Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/93
Other Adverse Events (participants affected / at risk) | 14/90 | 23/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Morphine (N=90) | Hydromorphone (N=93)
Nausea (Gastrointestinal disorders) | 4/46 | 5/48 — excludes patients who were nauseated or vomiting before baseline
Vomiting (Gastrointestinal disorders) | 1/46 | 0/48 — excludes patients who were nauseated or vomiting before baseline
Systolic blood pressure <90 mmHg (Vascular disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Respiratory rate <12 breaths/min (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oxygen saturation <90% (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oxygen saturation 90%-94% (Respiratory, thoracic and mediastinal disorders) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes